CLINICAL TRIAL: NCT01808599
Title: A Phase II Study of Chlorambucil in Combination With Subcutaneous Rituximab Followed by Maintenance Therapy With Subcutaneous Rituximab in Patients With Extranodal Marginal Zone B-cell Lymphoma of Mucosa Associated Lymphoid Tissue (MALT Lymphoma)
Brief Title: Phase II Study of Chlorambucil and Subcutaneous Rituximab in Patients With Extranodal MALT Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: International Extranodal Lymphoma Study Group (IELSG) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IELSG38
Record Dates: First submitted 2013-03-06; First posted 2013-03-11 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: MALT Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — Chlorambucil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chlorambucil, Rituximab i.v., Rituximab s.c. (Experimental): Chlorambucil 6 mg/m2 daily p.o for 42 consecutive days (weeks 1-6) in combination with intravenous Rituximab 375mg/m2 on days 1, 8, 15 and 22 (day 1 of weeks 1, 2, 3 and 4).
  Starting from d56, (month 3) patients will receive Chlorambucil 6 mg/m2 daily p.o for 14 consecutive days (d1-14) every 28 days for 4 cycles in combination with subcutaneous Rituximab 1400mg on day 1 of each 28-day cycle. Therefore subcutaneous Rituximab 1400mg every two months for 2 years (in total 12 injections).
  Interventions: Drug: Chlorambucil; Drug: Rituximab i.v.; Drug: Rituximab s.c.

INTERVENTIONS:
Drug: Chlorambucil
Drug: Rituximab i.v.
Drug: Rituximab s.c.

SUMMARY:
Single arm phase II study of Chlorambucil in combination with subcutaneous Rituximab followed by maintenance therapy with subcutaneous Rituximab in patients with histologically proven diagnosis of CD20-positive marginal zone B-cell lymphoma of MALT type arisen at any extranodal site, either de novo, or relapsed following local therapy (including surgery, radiotherapy and antibiotics for H. pylori-positive gastric lymphoma).

DETAILED DESCRIPTION:
The study consists in three parts. In Part A (induction phase I) patients will be treated with Chlorambucil 6 mg/m2 daily p.o for 42 consecutive days (weeks 1-6) in combination with intravenous Rituximab 375mg/m2 on day 1 week 1 followed by subcutaneous Rituximab 1400mg on days 8, 15 and 22 (day 1 of weeks 2, 3 and 4). After restaging (CT scan to be performed during weeks 7-8, i.e. between d42 and d55), responding patients (CR, CRu, PR) and those with stable disease will be treated in part B (induction phase II). In part B, starting from d56, (month 3) patients will receive Chlorambucil 6 mg/m2 daily p.o for 14 consecutive days (d1-14) every 28 days for 4 cycles in combination with subcutaneous Rituximab 1400mg on day 1 of each 28-day cycle. After restaging (CT scan to be performed at the end of month 6) responding patients and those with stable disease will be treated in part C. In Part C (maintenance phase) patients will be treated with subcutaneous Rituximab 1400mg every two months for 2 years (in total 12 injections). During maintenance phase, CT scans will be performed every 12 months and patients responding or with stable disease will stay on treatment for a total of two years as above reported.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven diagnosis of CD20-positive marginal zone B-cell lymphoma of MALT type either de novo, or relapsed following local therapy (including surgery, radiotherapy and antibiotics for H. pylori-positive gastric lymphoma) arisen at any extranodal site 1.1 The following patients with gastric MALT Lymphoma can be entered:

   * H. pylori-negative cases, either de novo (non pre-treated) or at relapse following local therapy (i.e., surgery, radiotherapy or antibiotics).
   * H. pylori-positive cases at diagnosis, who failed antibiotic therapy, including

     * Patients with clinical (endoscopic) and histological evidence of disease progression at any time post H. pylori eradication
     * Stable disease with persistent lymphoma at ≥ 1 year post H. pylori eradication
     * Relapse (without H. pylori re-infection), after a remission
     * Patients who failed either first line antibiotics or further local treatment (surgery or radiotherapy) 1.2 Similar consideration may be applied to patients with ocular adnexal lymphoma treated with antibiotics.
2. Measurable or evaluable disease. Measurable disease in at least two perpendicular dimensions on an imaging scan is defined as: lymph node or nodal mass bi-dimensional measurement with > 1.5 cm in longest transverse diameter or the short diameter must measure > 10 mm regardless of the longest transverse diameter.
3. Any stage (Ann Arbor I-IV) (see Appendix A)
4. Age ≥ 18
5. Life expectancy of at least 1 year
6. ECOG performance status 0-2 (see Appendix B)
7. Adequate bone marrow function (WBC >3.0x109/L, ANC >1.5x109/L, PLT >100x109/L), unless due to lymphoma involvement
8. Adequate kidney (serum creatinine <1,5x upper normal) and liver function (ASAT/ALAT <2,5 upper normal, total bilirubin <2,5x upper normal), unless due to lymphoma involvement
9. For women of childbearing potential only: negative serum pregnancy test done within 7 days prior to study drugs administration or within 14 days if with a confirmatory urine pregnancy test within 7 days prior to the first study drugs administration
10. Fertile male or female patients of childbearing potential and their partners must use two forms of contraception during the study and for at least 12 months after the last dose of subcutaneous rituximab.

    For appropriate methods of contraception considered acceptable, see Appendix C. Should a woman become pregnant or suspect she is pregnant while she or her partner are participating in this study and for 12 months after study participation, the patient should inform the treating physician immediately.

    Female patients of childbearing potential are defined as follows:
    * Pre-menopausal women (patients with regular menstruation, patients after menarche with amenorrhea or irregular cycles, patients using a contraceptive method that precludes withdrawal bleeding
    * Women who have had tubal ligation

    Female patients may be considered to NOT be of childbearing potential for the following reasons:
    * The patient has undergone total abdominal hysterectomy with bilateral salpingo-oophorectomy or bilateral oophorectomy
    * The patient is medically confirmed to be menopausal (no menstrual period) for 24 consecutive months
11. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Evidence of histologic transformation to a high grade lymphoma
2. Prior diagnosis of neoplasm within 5 years, except cervical intraepithelial neoplasia type 1 (CIN1) or localized non-melanomatous skin cancer
3. Prior chemotherapy
4. Prior immunotherapy with any anti-CD20 monoclonal antibody
5. Prior radiotherapy in the last 6 weeks
6. Use of corticosteroids during the last 28 days, unless prednisone chronically administered at a dose <20 mg/day for indications other than lymphoma or lymphoma-related symptoms
7. Evidence of clinically significant cardiac disease, as defined by history of symptomatic ventricular arrhythmias, congestive heart failure or myocardial infarction within 12 months before study entry
8. Evidence of symptomatic central nervous system (CNS) disease
9. Evidence of active opportunistic infections
10. Known HIV infection
11. Positive serology for Hepatitis B (HB) defined as a positive test for HBsAg. In addition, if negative for HBsAg but HBcAb positive (regardless of HBsAb status), a HBV DNA test will be performed and if positive the subject will be excluded
12. Positive serology for hepatitis C (HC) defined as a positive test for HCAb, confirmed by HC RIBA immunoblot assay on the same sample.
13. Pregnant or lactating status
14. Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
15. Fertile men or women of childbearing potential who do not agree to use a highly effective measure of contraception (such as oral contraceptives, intrauterine device or barrier method of contraception in conjunction with spermicidal jelly or surgically sterile) throughout the study and for at least 12 months after the last dose of subcutaneous rituximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2013-12; Primary Completion 2016-03 (Actual); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate | week 25

SECONDARY OUTCOMES:
Response Rate | week 25
  Response rate (Complete and partial remission rates) for all patients
Event-free-survival (EFS) | at 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele Zucca, MD, Principal Investigator — IOSI Oncology Institute of Southern Switzerland
Locations (38):
- France (14):
  - Créteil Hopital Henri Mondor, Créteil
  - Dijon CHU Hopital le Bocage, Dijon
  - Clermont Ferrand CHU Estaing, Estaing
  - Grenoble CHU Pontchaillou, Grenoble
  - Lille CHRU Hopital Claude Dieu, Lille
  - Pierre Bénite CHU Lyon Sud, Lyon
  - Marseille Paoli Calmettes, Marseille
  - Montpellier CHU Saint Eloi, Montpellier
  - Vandoeuvre lès Nancy CHU Brabois, Nancy
  - Nantes CHU Hotel Dieu, Nantes
  - Paris Hopital Saint Louis, Paris
  - Rennes CHU Pontchaillou, Rennes
  - Rouen Centre Henri Becquerel, Rouen
  - Tours CHU Bretonneau, Tours
- Italy (23):
  - AO SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Ancona, Ancona
  - Centro di Riferimento Oncologico di Aviano, Aviano
  - Biella Ospedale degli Infermi, Biella
  - Ematologia e CTMO Ospedale Bolzano, Bolzano
  - Ematologia Ospedale Businco (Cagliari), Cagliari
  - ARNAS Garibaldi Catania, Catania
  - Genova Ematologia I H San Martino, Genova
  - Azienda Sanitaria AUSL6 Livorno, Livorno
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola, Meldola
  - Istituto Nazionale dei Tumori, Milano, Milan
  - Milano Ospedale Policlinico, Milan
  - Nocera, Nocera Umbra
  - IOV Padova, Padua
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - UO Ematologia Ravenna, Ravenna
  - Arcispedale Santa Maria Nuova, Azienda Ospedaliera di Reggio Emilia, Reggio Emilia
  - Ospedale Infermi Ematologia Rimini, Rimini
  - IRCCS/CROB Rionero in Vulture, Rionero in Vulture
  - Istituto Regina Elena, Roma, IFO, Roma
  - SC Oncoematologia Terni, Terni
  - SC Ematologia Torino-Molinette, Torino
  - Torino Università, Ematologia 1, AO Città della Salute e della Scienza, Torino
- IOSI - Oncology Institute of Southern Switzerland, Bellinzona, Switzerland

REFERENCES:
- [Derived] Stathis A, Pirosa MC, Orsucci L, Feugier P, Tani M, Ghesquieres H, Musuraca G, Rossi FG, Merli F, Guieze R, Gyan E, Gini G, Marino D, Gressin R, Morschhauser F, Cavallo F, Palombi F, Conconi A, Tessoulin B, Tilly H, Zanni M, Cabras MG, Capochiani E, Califano C, Celli M, Pulsoni A, Angrilli F, Occhini U, Casasnovas RO, Cartron G, Devizzi L, Haioun C, Liberati AM, Houot R, Merli M, Pietrantuono G, Re F, Spina M, Landi F, Cavalli F, Bertoni F, Rossi D, Ielmini N, Borgo E, Luminari S, Zucca E, Thieblemont C. IELSG38: phase II trial of front-line chlorambucil plus subcutaneous rituximab induction and maintenance in mucosa-associated lymphoid tissue lymphoma. Haematologica. 2024 Aug 1;109(8):2564-2573. doi: 10.3324/haematol.2023.283918. PMID 38385243